CLINICAL TRIAL: NCT02948621
Title: Endoscopic Sleeve Gastroplasty
Acronym: Endosleeve
Status: Completed | Type: Observational
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Other Study IDs: 16-001-OBS
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Morbid Obesity
Keywords: Endoscopic sleeve gastroplasty; Excess weight loss; Quality of life
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic sleeve gastroplasty: Endoscopic sleeve gastroplasty is performed using a CE marked endoscopic suture device (Overstitch, Apollo Endosurgery, Austin, Tx. USA). Continuous stitches are placed to create a sleeve-shaped gastric path of 2 cm diameter to reduce stomach volume from the proximal antrum to the oeso-gastric junction.
  Interventions: Procedure: Endoscopic sleeve gastroplasty

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty — Endoscopic sleeve gastroplasty is performed using a CE marked endoscopic suture device (Overstitch, Apollo Endosurgery, Austin, Tx. USA). Continuous stitches are placed to create a sleeve-shaped gastric path of 2 cm diameter to reduce stomach volume from the proximal antrum to the oeso-gastric junction.

SUMMARY:
The endoscopic sleeve gastroplasty allows stomach size reduction through an endoluminal suture approach without any incision. It could reduce the complications associated with current surgical techniques while obtaining the target gastric restriction, weight loss, comorbidities and quality of life improvement.

The primary objective of this study is to assess weight loss after endoscopic sleeve gastroplasty in patients with morbid obesity.

DETAILED DESCRIPTION:
Gastric restriction is one of the fundamental principles of gastric bypass and gastric banding. Nowadays, practitioners have the possibility to reduce stomach size by merging tissues through an endoscopic endoluminal suture approach without any incision. This could reduce the complications associated with current surgical techniques while obtaining the target gastric restriction, weight loss, comorbidities and quality of life improvement.

The primary objective of this study is to assess weight loss after endoscopic sleeve gastroplasty in patients with morbid obesity according to the technique described in the literature: reduction of the gastric pouch into a sleeve structure by modification of the stomach greater curvature thanks to a plication.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old and < 60 years old
* Patient with morbid obesity for at least 2 years
* Patient who failed medical and diet treatment of obesity
* Patient with no contraindication to anesthesia
* Patient able to understand the study and to provide informed consent.

Exclusion Criteria:

* Patient with inflammatory, tumoral or bad quality tissues at endoscopy
* Patient with a history of gastro-intestinal inflammatory disease, stenosis or intestinal adhesions, kidney or liver failure, chronic pancreatic disease
* Patient with a history and/or signs and/or symptoms of gastroduodenal ulcerous disease and/or progressive gastroduodenal ulcerous disease
* Patient with an oesophageal pathology as Zenker's diverticulum, peptic oesophagitis stage 3-4, oesophageal stenosis, Barrett syndrome, oesophageal cancer, dysphagia, achalasia
* Patient with previous bariatric, gastric or oesophageal surgery, intestinal obstruction, portal hypertension, gastro-intestinal tumors, oesophageal or gastric varices, gastroparesis
* Patient with a severe coagulopathy (prothrombin time > 3 seconds or thrombocytic count < 50 000/mm3) or treated with heparin, coumadin, warfarin or any other anticoagulants and drugs preventing coagulation or platelet aggregation, except aspirin and nonsteroidal anti-inflammatory drugs
* Pregnancy, breastfeeding or woman without contraception
* Patient with a congestive heart failure, arrhythmia or unstable coronary heart disease
* Patient using or having used diet drugs within the last 30 days or intending to use them during study follow-up
* Patient under drug treatment within the last 3 months known to induce weight gain
* Patient with eating disorders or uncontrolled, poorly controlled or suspected psychiatric disease
* Patient in a poor condition according to investigator
* Patient in exclusion period (determined by a previous study or in progress)
* Patient with significative weight loss between date of enrollment in the study and date of procedure
* Patient with a systemic infection the day of procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients over 18 years old requiring a treatment for morbid obesity.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
Excess weight loss | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
Body mass index variation | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure

SECONDARY OUTCOMES:
Procedure reproducibility | 7 days, 1 - 3 - 6 - 9 and 12 months after procedure
  Absence of adverse event within 12 months after procedure.
Comorbidities improvement | 7 days, 1 - 3 - 6 - 9 - 12 - 18 and 24 months after procedure
  Improvement of hyperlipidemia, arterial hypertension, diabetes, reflux, osteoarticular disorders compared with preoperative data.
Quality of life improvement | 3 - 12 - 18 and 24 months after procedure
  Improvement of quality of life assessed by Moorehead-Ardelt Quality of life II questionnaire and Gastro-intestinal Quality of Life Index questionnaire.
Modification in the feeling of satiety | 1 - 3 - 6 - 12 - 18 and 24 months after procedure
  Satiety assessed by Three Factors Eating Questionnaire - R18.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Perretta, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil de Strasbourg; Michel Vix, MD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez-Nava G, Galvao MP, da Bautista-Castano I, Jimenez A, De Grado T, Fernandez-Corbelle JP. Endoscopic sleeve gastroplasty for the treatment of obesity. Endoscopy. 2015 May;47(5):449-52. doi: 10.1055/s-0034-1390766. Epub 2014 Nov 7. PMID 25380508
- [Background] Lopez-Nava G, Galvao MP, Bautista-Castano I, Jimenez-Banos A, Fernandez-Corbelle JP. Endoscopic Sleeve Gastroplasty: How I Do It? Obes Surg. 2015 Aug;25(8):1534-8. doi: 10.1007/s11695-015-1714-7. PMID 26003549
- [Background] Lopez-Nava G, Galvao M, Bautista-Castano I, Fernandez-Corbelle JP, Trell M. Endoscopic sleeve gastroplasty with 1-year follow-up: factors predictive of success. Endosc Int Open. 2016 Feb;4(2):E222-7. doi: 10.1055/s-0041-110771. Epub 2016 Jan 15. PMID 26878054
- [Background] Sharaiha RZ, Kedia P, Kumta N, DeFilippis EM, Gaidhane M, Shukla A, Aronne LJ, Kahaleh M. Initial experience with endoscopic sleeve gastroplasty: technical success and reproducibility in the bariatric population. Endoscopy. 2015 Feb;47(2):164-6. doi: 10.1055/s-0034-1390773. Epub 2014 Nov 7. PMID 25380510
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556